CLINICAL TRIAL: NCT07154680
Title: Ophthalmic Diseases and AI: an Parallel Comparison RCT Study
Brief Title: Ophthalmic Diseases and AI: an RCT Study
Status: Completed | Type: Observational
Sponsor: North Sichuan Medical College (Other)
Collaborators: Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Principal Investigator, Zining Luo, Principal Investigator, North Sichuan Medical College
Other Study IDs: 2765326471-2024-1
Record Dates: First submitted 2024-12-29; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Large Language Model Diagnostics Group
  Interventions: Diagnostic Test: GPT-4o mini;Claude 3 Haiku;Gemini 1.5 Flash;Llama 3.1 7OB;GPT-4o;Claude 3.5 Sonnet;Gemini 1.5 Pro;Llama 3.1 4O5B
- Large Language Model Medical Assistance Group
  Interventions: Diagnostic Test: GPT-4o mini;Claude 3 Haiku;Gemini 1.5 Flash;Llama 3.1 7OB;GPT-4o;Claude 3.5 Sonnet;Gemini 1.5 Pro;Llama 3.1 4O5B
- Large Language Model Medical Explanation Team
  Interventions: Diagnostic Test: GPT-4o mini;Claude 3 Haiku;Gemini 1.5 Flash;Llama 3.1 7OB;GPT-4o;Claude 3.5 Sonnet;Gemini 1.5 Pro;Llama 3.1 4O5B

INTERVENTIONS:
Diagnostic Test: GPT-4o mini;Claude 3 Haiku;Gemini 1.5 Flash;Llama 3.1 7OB;GPT-4o;Claude 3.5 Sonnet;Gemini 1.5 Pro;Llama 3.1 4O5B — Input all the patient's information into the large language model and process it using a pre-defined prompt.

SUMMARY:
Ophthalmic diseases are a major category of conditions affecting visual health, including but not limited to cataracts, glaucoma, retinal and choroidal diseases, and refractive errors (such as myopia, hyperopia, and astigmatism). With the advancement of technology, artificial intelligence (AI) is being increasingly applied in the field of ophthalmology. This clinical trial aims to evaluate the potential of large language models (LLMs) in ophthalmology.

The main questions to be addressed are:

1. Assessing the effectiveness of large language models (LLMs) in the diagnosis and treatment of ophthalmic diseases: Through randomized controlled trials (RCTs), evaluate the diagnostic and treatment effectiveness of LLMs in the field of ophthalmic diseases, exploring their potential to improve the quality and efficiency of ophthalmic care.
2. Investigating the role of LLMs in medical consultations: Explore the role and effectiveness of LLMs in medical consultations for ophthalmic diseases, including their ability to provide medical advice, explain diagnostic results, and help patients understand treatment plans.
3. Examining the ability of LLMs to adhere to ethical standards: Study how to ensure that LLMs comply with ethical standards and moral principles in ophthalmic medical consultations, safeguarding patient privacy and rights.
4. Providing new technological support for the field of ophthalmology: Through research on the application of LLMs in ophthalmic diseases, offer new technological support and innovations to enhance the quality and efficiency of ophthalmic care.
5. Exploring the differences between LLMs and ophthalmologists: By utilizing multiple large language models, compare the differences between LLMs and ophthalmologists in diagnostic outcomes, case analysis processes, and patient experiences during diagnosis and treatment.
6. Evaluating the effectiveness of LLMs in ophthalmic diseases: Collect patient complaints, fundus images, doctors' diagnoses, and diagnosis times from offline doctor consultations, as well as gather AI-generated medical advice, diagnostic efficiency, and diagnostic accuracy online. Ultimately, conduct comprehensive data analysis to determine the feasibility and effectiveness of LLMs in diagnosing and treating ophthalmic diseases.

ELIGIBILITY:
Inclusion Criteria:

* There are patient complaints

Exclusion Criteria:

* No patient complaints

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients going to the hospital for regular eye check-ups
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Large Language Model Diagnostics | 1 week
  The accuracy of the large language model in diagnosing eye diseases

SECONDARY OUTCOMES:
Large Language Model Medical Assistance | 1 week
  The time of diagnosis of eye diseases and other information of the large language model

OTHER OUTCOMES:
Large Language Model Medical Explanation | 1 week
  Large language models diagnose the process of eye disease, attitude to patients, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Afﬁliated Hospital of North Sichuan Medical College, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code